CLINICAL TRIAL: NCT03345537
Title: Observational Prospective Multicentered Study Evaluating Initial Clinical Presentation of Inflammatory Optic Neuritis (ON) Associated or Not With Autoantibodies Anti- Myelin-oligodendrocyte-glycoprotein (MOG-Ab)
Brief Title: Initial Clinical Presentation of Inflammatory Optic Neuritis Associated or Not With Autoantibodies Anti-Myelin-oligodendrocyte-glycoprotein
Acronym: MOG
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0250
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Optic Neuritis
Keywords: Inflammatory; Optic neuritis; autoantibodies anti MOG
MeSH Terms: conditions — Optic Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample (5mL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non interventional study — Non interventional study - only data collected and one blood sample additional

SUMMARY:
In eight ophthalmic units, the investigator will include all inflammatory optic neuritis (ON) during acute phase and rank them in two groups: 1/ ON with autoantibodies anti-myelin-oligodendrocyte-glycoprotein (ON MOG+) 2/ ON MOG-. The investigators will measure incidence of MOG-Ab in our prospective population of inflammatory ON. Then the investigator will compare clinical and radiological presentation of ON MOG+ versus ON MOG-.

DETAILED DESCRIPTION:
Optic neuritis (ON) have a broad clinical spectrum ranging from a single episode (clinically isolated ON) to demyelinating diseases such as multiple sclerosis (MS), Chronic Relapsing Inflammatory Optic Neuritis (CRION), acute demyelination encephalomyelitis (ADEM), neuromyelitis optica (NMO) and neuromyelitis optica spectrum disorder (NMOSD). Myelin oligodendrocyte glycoprotein (MOG) is a myelin antigen exclusively expressed on the surface of oligodendrocytes and myelin in the central nervous system (CNS). MOG-Ab are associated with demyelinating diseases with a good specificity. Using cell-based assays, MOG-Ab were rarely found in healthy control and other neurological inflammatory disease. They were mostly identified in subgroups of NMO/NMOSD seronegative to auto antibodies against Aquaporin 4 (anti-AQP4): 8-39%, but also in MS (0-28%) ADEM and idiopathic ON. ON MOG + have a specific clinical presentation compare with ON associated with multiple sclerosis (SEP): older patient, less female preponderance, more often bilateral, more often optic disc swelling, worse initial visual loss, much more often recurrent with severe sequelae. ON MOG+ are more similar to ON associated with NMOSD AQP4+ which have some particularities: similar age, clear female preponderance, less optic disc swelling, more severe initial visual loss and visual sequelae. No prospective study has measured incidence of

MOG-Ab in population of Inflammatory ON. And no prospective study has ever compared ON MOG+ with all others inflammatory ON. The purpose of our study is to measure incidence of MOG-Ab in population of acute inflammatory ON. All consenting adults with suspicion of ON followed in the 8 ophthalmic units who participate will be screened. They will have, as usual, clinical follow-up, blood test with MOG-Ab research, encephalic and optic nerves MRI, and steroid treatment if necessary. At the end of the acute phase, all patients diagnosed with inflammatory ON will be included and rank in 2 groups: 1/ ON with MOG-Ab (ON MOG+) 2/ ON without MOG-Ab (ON MOG-). Clinical data will be register at this inclusion visit. There will be no additional visit and no intervention. After measuring incidence of MOG-Ab, the investigator will compare clinical and radiological data of ON MOG+ and ON MOG-.

ELIGIBILITY:
Inclusion Criteria:

* legally adult patient
* acute inflammatory optic neuritis
* consent

Exclusion Criteria:

* Patient under tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phe patients included will be mostly young adults between 18 and 40 years old, consultant in the ophthalmology department of the University Hospital of Nantes for an inflammatory optic neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of anti-Myelin-oligodendrocyte-glycoprotein (MOG-ab) | the day of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Lebranchu, Dr, Principal Investigator — Nantes University Hospital
Locations (8):
- France (8):
  - Chu Angers, Angers
  - Ch Challans, Challans
  - Ch Cholet, Cholet
  - Chd La Roche Sur Yon, La Roche-sur-Yon
  - Ch Laval, Laval
  - Chr Le Mans, Le Mans
  - CHU Nantes, Nantes
  - Ch Saint Nazaire, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramanathan S, Dale RC, Brilot F. Anti-MOG antibody: The history, clinical phenotype, and pathogenicity of a serum biomarker for demyelination. Autoimmun Rev. 2016 Apr;15(4):307-24. doi: 10.1016/j.autrev.2015.12.004. Epub 2015 Dec 17. PMID 26708342
- [Background] Akaishi T, Nakashima I, Takeshita T, Kaneko K, Mugikura S, Sato DK, Takahashi T, Nakazawa T, Aoki M, Fujihara K. Different etiologies and prognoses of optic neuritis in demyelinating diseases. J Neuroimmunol. 2016 Oct 15;299:152-157. doi: 10.1016/j.jneuroim.2016.09.007. Epub 2016 Sep 14. PMID 27725114
- [Background] Ramanathan S, Reddel SW, Henderson A, Parratt JD, Barnett M, Gatt PN, Merheb V, Kumaran RY, Pathmanandavel K, Sinmaz N, Ghadiri M, Yiannikas C, Vucic S, Stewart G, Bleasel AF, Booth D, Fung VS, Dale RC, Brilot F. Antibodies to myelin oligodendrocyte glycoprotein in bilateral and recurrent optic neuritis. Neurol Neuroimmunol Neuroinflamm. 2014 Oct 29;1(4):e40. doi: 10.1212/NXI.0000000000000040. eCollection 2014 Dec. PMID 25364774
- [Background] Havla J, Kumpfel T, Schinner R, Spadaro M, Schuh E, Meinl E, Hohlfeld R, Outteryck O. Myelin-oligodendrocyte-glycoprotein (MOG) autoantibodies as potential markers of severe optic neuritis and subclinical retinal axonal degeneration. J Neurol. 2017 Jan;264(1):139-151. doi: 10.1007/s00415-016-8333-7. Epub 2016 Nov 14. PMID 27844165
- [Background] Sato DK, Callegaro D, Lana-Peixoto MA, Waters PJ, de Haidar Jorge FM, Takahashi T, Nakashima I, Apostolos-Pereira SL, Talim N, Simm RF, Lino AM, Misu T, Leite MI, Aoki M, Fujihara K. Distinction between MOG antibody-positive and AQP4 antibody-positive NMO spectrum disorders. Neurology. 2014 Feb 11;82(6):474-81. doi: 10.1212/WNL.0000000000000101. Epub 2014 Jan 10. PMID 24415568
- [Background] Jarius S, Ruprecht K, Kleiter I, Borisow N, Asgari N, Pitarokoili K, Pache F, Stich O, Beume LA, Hummert MW, Ringelstein M, Trebst C, Winkelmann A, Schwarz A, Buttmann M, Zimmermann H, Kuchling J, Franciotta D, Capobianco M, Siebert E, Lukas C, Korporal-Kuhnke M, Haas J, Fechner K, Brandt AU, Schanda K, Aktas O, Paul F, Reindl M, Wildemann B; in cooperation with the Neuromyelitis Optica Study Group (NEMOS). MOG-IgG in NMO and related disorders: a multicenter study of 50 patients. Part 2: Epidemiology, clinical presentation, radiological and laboratory features, treatment responses, and long-term outcome. J Neuroinflammation. 2016 Sep 27;13(1):280. doi: 10.1186/s12974-016-0718-0. PMID 27793206
- [Background] Hoftberger R, Sepulveda M, Armangue T, Blanco Y, Rostasy K, Calvo AC, Olascoaga J, Ramio-Torrenta L, Reindl M, Benito-Leon J, Casanova B, Arrambide G, Sabater L, Graus F, Dalmau J, Saiz A. Antibodies to MOG and AQP4 in adults with neuromyelitis optica and suspected limited forms of the disease. Mult Scler. 2015 Jun;21(7):866-874. doi: 10.1177/1352458514555785. Epub 2014 Oct 24. PMID 25344373
- [Background] The clinical profile of optic neuritis. Experience of the Optic Neuritis Treatment Trial. Optic Neuritis Study Group. Arch Ophthalmol. 1991 Dec;109(12):1673-8. doi: 10.1001/archopht.1991.01080120057025. PMID 1841573
- [Background] Stiebel-Kalish H, Lotan I, Brody J, Chodick G, Bialer O, Marignier R, Bach M, Hellmann MA. Retinal Nerve Fiber Layer May Be Better Preserved in MOG-IgG versus AQP4-IgG Optic Neuritis: A Cohort Study. PLoS One. 2017 Jan 26;12(1):e0170847. doi: 10.1371/journal.pone.0170847. eCollection 2017. PMID 28125740
- [Background] Beck RW, Cleary PA, Anderson MM Jr, Keltner JL, Shults WT, Kaufman DI, Buckley EG, Corbett JJ, Kupersmith MJ, Miller NR, et al. A randomized, controlled trial of corticosteroids in the treatment of acute optic neuritis. The Optic Neuritis Study Group. N Engl J Med. 1992 Feb 27;326(9):581-8. doi: 10.1056/NEJM199202273260901. PMID 1734247
- [Background] Elsone L, Panicker J, Mutch K, Boggild M, Appleton R, Jacob A. Role of intravenous immunoglobulin in the treatment of acute relapses of neuromyelitis optica: experience in 10 patients. Mult Scler. 2014 Apr;20(4):501-4. doi: 10.1177/1352458513495938. Epub 2013 Aug 28. PMID 23986097
- [Background] Optic Neuritis Study Group. Visual function 15 years after optic neuritis: a final follow-up report from the Optic Neuritis Treatment Trial. Ophthalmology. 2008 Jun;115(6):1079-1082.e5. doi: 10.1016/j.ophtha.2007.08.004. Epub 2007 Nov 5. PMID 17976727
- [Background] Garcia-Martin E, Ara JR, Martin J, Almarcegui C, Dolz I, Vilades E, Gil-Arribas L, Fernandez FJ, Polo V, Larrosa JM, Pablo LE, Satue M. Retinal and Optic Nerve Degeneration in Patients with Multiple Sclerosis Followed up for 5 Years. Ophthalmology. 2017 May;124(5):688-696. doi: 10.1016/j.ophtha.2017.01.005. Epub 2017 Feb 7. PMID 28187977
- [Background] Beck RW, Gal RL, Bhatti MT, Brodsky MC, Buckley EG, Chrousos GA, Corbett J, Eggenberger E, Goodwin JA, Katz B, Kaufman DI, Keltner JL, Kupersmith MJ, Miller NR, Moke PS, Nazarian S, Orengo-Nania S, Savino PJ, Shults WT, Smith CH, Trobe JD, Wall M, Xing D; Optic Neuritis Study Group. Visual function more than 10 years after optic neuritis: experience of the optic neuritis treatment trial. Am J Ophthalmol. 2004 Jan;137(1):77-83. doi: 10.1016/s0002-9394(03)00862-6. PMID 14700647
- [Background] Pache F, Zimmermann H, Mikolajczak J, Schumacher S, Lacheta A, Oertel FC, Bellmann-Strobl J, Jarius S, Wildemann B, Reindl M, Waldman A, Soelberg K, Asgari N, Ringelstein M, Aktas O, Gross N, Buttmann M, Ach T, Ruprecht K, Paul F, Brandt AU; in cooperation with the Neuromyelitis Optica Study Group (NEMOS). MOG-IgG in NMO and related disorders: a multicenter study of 50 patients. Part 4: Afferent visual system damage after optic neuritis in MOG-IgG-seropositive versus AQP4-IgG-seropositive patients. J Neuroinflammation. 2016 Nov 1;13(1):282. doi: 10.1186/s12974-016-0720-6. PMID 27802824